CLINICAL TRIAL: NCT01427920
Title: A 20 Week Randomised, Multinational, Open Labelled, 2 Armed, Parallel Group Comparison of Twice Daily Subject Driven Titration of Biphasic Insulin Aspart (BIAsp) 30 Versus Twice Daily Investigator-driven Titration of Biphasic Insulin Aspart (BIAsp) 30 Both in Combination With Metformin in Subjects With Type 2 Diabetes Inadequately Controlled on Basal Insulin Analogues
Brief Title: Comparison of Biphasic Insulin Aspart 30 Individually Adjusted by the Subject and the Trial Physician, Both Combined With Metformin in Subjects With Type 2 Diabetes
Acronym: SimpleMix™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3878; 2010-024303-27 (EudraCT Number); U1111-1118-4096 (Other: WHO)
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2013-09-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subject-driven titration BIAsp 30 (BID) + metformin (Experimental): The subjects performed the titration of BIAsp 30 dose.
  Interventions: Drug: biphasic insulin aspart 30
- Investigator-driven titration BIAsp 30 (BID) + metformin (Active Comparator): The investigator performed the titration of BIAsp 30 dose.
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Administered subcutaneously (under the skin) using FlexPen® twice daily for 20 weeks. Directions for use were given to each subject at each dispensing visit. Subjects continued on their pre-trial metformin dose. Any previous basal insulin analogue and OAD (oral anti-diabetes drug) treatments (except for metformin) were discontinued.

SUMMARY:
This trial was conducted in Asia, Europe and South America. The aim of this trial was to confirm efficacy of subject driven titration (individually adjusted) of biphasic insulin aspart 30 (BIAsp 30) twice daily in terms of glycaemic control assessed by change in glycosylated haemoglobin (HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for a minimum of 12 months prior to Visit 1 (screening)
* Currently treated with a basal insulin analogue for at least 3 months prior to Visit 1 (screening)
* Stable treatment (no change in dose or regimen) with a total daily dose of at least 1500 mg metformin or maximum tolerated dose (minimum 1000 mg) ± additional OAD treatment. The metformin treatment must have been stable for at least 2 months prior to Visit 1 (screening)
* HbA1c higher or equal to 7.0% and below or equal to 10.0% (one re-test within one week of screening visit was allowed. The last sample was to be conclusive)
* Body Mass Index (BMI) below or equal to 40.0 kg/m^2
* Able and willing to eat at least 2 main meals each day during the trial
* Able and willing to adhere to the protocol including compliance with performance of self measured plasma glucose (SMPG), injection regimen and titrating themselves according to the protocol
* Experience in performing self measured plasma glucose (SMPG)

Exclusion Criteria:

* Treatment with any thiazolidinedione (TZD) and glucagon-like peptide-1 (GLP-1) receptor agonists or pramlintide within the last 3 months prior to Visit 1 (screening)
* Impaired hepatic function defined as alanine aminotransferase (ALAT) above or equal to 2.5 times upper referenced limit (one re-test within one week of screening visit was allowed. The last sample was to be conclusive)
* Impaired kidney function with serum creatinine above or equal to 133 micromol/L (1.5 mg/dL) for males and above or equal to 124 micromol/L (1.4 mg/dL) for females (one re-test within one week of screening visit was allowed. The last sample was to be conclusive)
* Cardiac problems or uncontrolled treated/untreated severe hypertension (defined as systolic blood pressure higher or equal to 180 mmHg and/or diastolic blood pressure higher or equal to 100 mmHg)
* Previous use of pre-mixed insulin products (pre-mixed insulin analogues or pre-mixed human preparations) or bolus insulin. Previous use of pre-mixed or bolus insulin products was allowed only in case of hospitalisation or a severe condition requiring intermittent use of pre-mixed or bolus insulin products for less than 14 consecutive days, but not during the last 3 months prior to screening visit (Visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (39):
- Argentina (3):
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Chacabuco
  - Novo Nordisk Investigational Site, Córdoba
- China (6):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Lanzhou, Gansu
  - Novo Nordisk Investigational Site, Zhengzhou, Henan
  - Novo Nordisk Investigational Site, Dalian, Liaoning
  - Novo Nordisk Investigational Site, Tianjin
- India (8):
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Belagavi, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, New Delhi, New Delhi
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Thriruvananthapuram
- Poland (8):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lubin
  - Novo Nordisk Investigational Site, Ruda Śląska
  - Novo Nordisk Investigational Site, Sopot
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Spain (7):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Centelles (Barcelona)
  - Novo Nordisk Investigational Site, La Roca Del Vallés (Barcelona)
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Vic (Barcelona)
- United Kingdom (7):
  - Novo Nordisk Investigational Site, Doncaster
  - Novo Nordisk Investigational Site, Ipswich
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Northwood
  - Novo Nordisk Investigational Site, Reading
  - Novo Nordisk Investigational Site, Scunthorpe
  - Novo Nordisk Investigational Site, Wirral, Merseyside

REFERENCES:
- [Result] Gao Y, Luquez C, Lynggaard H, Andersen H, Saboo B. The SimpleMix study with biphasic insulin aspart 30: a randomized controlled trial investigating patient-driven titration versus investigator-driven titration. Curr Med Res Opin. 2014 Dec;30(12):2483-92. doi: 10.1185/03007995.2014.960512. Epub 2014 Sep 29. PMID 25180608
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 33 sites in 5 countries enrolled subjects.
Groups:
- Subject-driven: The subjects performed the titration of biphasic insulin aspart 30 (BIAsp 30) dose and administered subcutaneously (under the skin) using FlexPen® twice daily for 20 weeks. The starting dose of BIAsp 30 was subject's previous basal insulin analogue dose split into two equal daily doses, immediately before breakfast and immediately before dinner. Directions for use were given to each subject at each dispensing visit. Subjects continued on their pre-trial metformin dose. Any previous basal insulin analogue and OAD (oral anti-diabetes drug) treatments (except for metformin) were discontinued. Metformin was allowed to be continued at the pre-trial dose with a total daily dose of at least 1500 mg or maximum tolerated dose (minimum 1000 mg) as prior to randomisation.
- Investigator-driven: The investigator performed the titration of biphasic insulin aspart 30 (BIAsp 30) dose and administered subcutaneously (under the skin) using FlexPen® twice daily for 20 weeks. The starting dose of BIAsp 30 was subject's previous basal insulin analogue dose split into two equal daily doses, immediately before breakfast and immediately before dinner. Directions for use were given to each subject at each dispensing visit. Subjects continued on their pre-trial metformin dose. Any previous basal insulin analogue and OAD (oral anti-diabetes drug) treatments (except for metformin) were discontinued. Metformin was allowed to be continued at the pre-trial dose with a total daily dose of at least 1500 mg or maximum tolerated dose (minimum 1000 mg) as prior to randomisation.
Period: Overall Study
Arm/Group | Subject-driven | Investigator-driven
Started | 174 | 174
Exposed | 174 | 173 (One subject withdrew prior to exposure to trial drug)
Completed | 165 | 157
Not Completed | 9 | 17
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal Criteria | 4 | 4
Not completed — Unclassified | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subject-driven | Investigator-driven | Total
Number analyzed (Participants) | 174 | 174 | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (9.8) | 58.0 (9.5) | 58.5 (9.6)
Gender [Count of Participants; unit: Participants]
  Female | 83 | 87 | 170
  Male | 91 | 87 | 178
Body Weight [Mean (Standard Deviation); unit: kg] | 81.0 (16.2) | 78.0 (15.0) | 79.5 (15.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (4.8) | 29.2 (4.7) | 29.4 (4.7)
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.9) | 8.3 (0.9) | 8.3 (0.9)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mmol/L] | 9.1 (2.7) | 8.8 (2.8) | 9.0 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin) - FAS
Description: Estimated mean change from baseline in HbA1c after 20 Weeks of treatment in full analysis set (FAS).
Time Frame: Week 0, week 20
Population: Full analysis set (FAS) - analysis included endpoint derived after 20 Weeks of treatment and missing data was imputed using last observation carried forward (LOCF) where any post-baseline measurements were available. 13 subjects did not contribute to the statistical analysis after Week 20.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Subject-driven | Investigator-driven
Number analyzed (Participants) | 169 | 166
percentage of glycosylated haemoglobin | -0.72 (0.08) | -0.97 (0.08)
Statistical Analysis 1: Comparison: Subject-driven vs Investigator-driven; FAS; Test type: Non-Inferiority or Equivalence — Non-inferiority for subject-driven vs. investigator driven titration would be concluded if the upper bound of the two-sided 95% CI was below or equal to 0.4%; Regression, Linear; Model includes treatment, strata and region as factors and relevant baseline HbA1c as covariate; Estimated treatment difference, Mean = 0.25, 95% CI [0.04 to 0.46]

2. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin) - PP
Description: Estimated mean change from baseline in HbA1c after 20 Weeks of treatment in per protocol (PP) analysis set.
Time Frame: Week 0, week 20
Population: Per protocol (PP) analysis set - analysis included subjects exposed to BIAsp 30 for more than 12 weeks without any major protocol violations. 24 subjects did not contribute to the statistical analysis after Week 20.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Subject-driven | Investigator-driven
Number analyzed (Participants) | 164 | 160
percentage of glycosylated haemoglobin | -0.71 (0.08) | -0.98 (0.08)
Statistical Analysis 1: Comparison: Subject-driven vs Investigator-driven; PP; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Regression, Linear; Model includes treatment, strata and region as factors and relevant baseline HbA1c as covariate; Estimated treatment difference, Mean = 0.26, 95% CI [0.05 to 0.48]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) (Central Laboratory Values)
Description: Estimated mean change from baseline in FPG after 20 Weeks of treatment
Time Frame: Week 0, week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Subject-driven | Investigator-driven
Number analyzed (Participants) | 169 | 166
mmol/L | -0.94 (0.21) | -1.07 (0.22)
Statistical Analysis 1: Comparison: Subject-driven vs Investigator-driven; H0: D = 0.0% against HA: D ≠ 0.0%, where D is the mean treatment difference (subject-driven titration minus investigator-driven titration); Test type: Superiority or Other; p = 0.659, Regression, Linear; Model includes treatment, strata and region as factors and relevant baseline FPG as covariate; Estimated treatment difference, Mean = 0.13, 95% CI [-0.44 to 0.69]

4. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes
Description: A hypoglycaemic episode was defined as treatment emergent if the onset of the episode was on or after the first day of trial product, and no later than one day after product administration. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to week 20
Population: Safety analysis set included all subjects who received at least one dose of BIAsp 30. One subject did not contribute to data.
Measure: Number; unit: episodes
Arm/Group | Subject-driven | Investigator-driven
Number analyzed (Participants) | 174 | 173
episodes | 638 | 766

5. Secondary Outcome: Patient Reported Outcomes Evaluated: Treatment-Related Impact Measures for Diabetes (TRIM-D) - Total Score
Description: From the 20 TRIM-D items, an overall score was derived. The scores were transformed to a 0 - 100 scale with higher scores indicating a better health state.
Time Frame: Week 0
Population: Full analysis set (FAS) - analysis included endpoint derived after 20 weeks of treatment and missing data was imputed using last observation carried forward (LOCF) where any post-baseline measurements were available. 10 subjects did not contribute to data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subject-driven | Investigator-driven
Number analyzed (Participants) | 169 | 169
scores on a scale | 67.2 (14.7) | 70.0 (15.3)

6. Secondary Outcome: Patient Reported Outcomes Evaluated: Treatment-Related Impact Measures for Diabetes (TRIM-D) - Total Score
Description: as for outcome 5
Time Frame: Week 4
Population: Full analysis set (FAS) - analysis included endpoint derived after 20 weeks of treatment and missing data was imputed using last observation carried forward (LOCF) where any post-baseline measurements were available. 20 subjects did not contribute to data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subject-driven | Investigator-driven
Number analyzed (Participants) | 165 | 163
scores on a scale | 71.0 (13.1) | 71.8 (14.4)

7. Secondary Outcome: Patient Reported Outcomes Evaluated: Treatment-Related Impact Measures for Diabetes (TRIM-D) - Total Score
Description: as for outcome 5
Time Frame: Week 20
Population: Full analysis set (FAS) - analysis included endpoint derived after 20 weeks of treatment and missing data was imputed using last observation carried forward (LOCF) where any post-baseline measurements were available. 17 subjects did not contribute to data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subject-driven | Investigator-driven
Number analyzed (Participants) | 167 | 164
scores on a scale | 73.9 (13.6) | 74.0 (15.4)

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the time of consent until 20 weeks of treatment, and if needed, were followed-up after the final visit.
Description: Safety analysis set included all subjects receiving at least one dose of BIAsp 30. Subjects in the safety set contributed to the evaluation "as treated".
Arm/Group | Subject-driven | Investigator-driven
Serious Adverse Events (participants affected / at risk) | 2/174 | 3/173
Other Adverse Events (participants affected / at risk) | 0/174 | 0/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject-driven (N=174) | Investigator-driven (N=173)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Novo Nordisk reserves the right to prior review of such publications and to ask for delay of publication of individual site results until after the primary manuscript is accepted for publication.